CLINICAL TRIAL: NCT01183585
Title: A Single Center, Open-label, Fixed Sequence, Two-period Study to Investigate the Effect of RO4917838 on the Pharmacokinetics of Rosuvastatin in Healthy Volunteers
Brief Title: A Study of RO4917838 With Rosuvastatin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP25262; 2010-020082-24
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Rosuvastatin Calcium

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RO4917838 and Rosuvastatin

INTERVENTIONS:
Drug: RO4917838 and Rosuvastatin — multiple oral doses of RO4917838 and single oral dose of Rosuvastatin

SUMMARY:
This single centre, open-label study will investigate the effect of RO4917838 on the pharmacokinetics of Rosuvastatin, a frequently co-prescribed drug in healthy volunteers. Healthy volunteers will receive multiple oral doses of RO4917838 and single oral dose of Rosuvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers, 18 to 65 years of age
* A body mass index (BMI) between 18 to 30 kg/m2

Exclusion Criteria:

* History of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardio-vascular, endocrinological, hematological or allergic disease, metabolic disorder, cancer or cirrhosis (Gilbert's Syndrome is allowed)
* Diseases or medical conditions that are capable of altering the absorption, metabolism or elimination of drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine the effect of multiple doses of RO4917838 on single-dose pharmacokinetics of Rosuvastatin | 30 days

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of single-dose Rosuvastatin and multiple-dose RO4917838 alone and in combination | 30 days
To explore the effect of single-dose Rosuvastatin on steady-state pharmacokinetics of RO4917838 | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Strasbourg, France